CLINICAL TRIAL: NCT01282320
Title: WHAT - Effectiveness of Physical Activity for Treatment of Hot Flushes Among Postmenopausal Women. A Randomized Controlled Pragmatic Pilot Study
Brief Title: WHAT (Women, Hot-flashes, Activity, Trial) - Physical Activity for Treatment of Hot Flushes Among Postmenopausal Women
Acronym: WHAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: University of Tromso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REK2009/1429
Record Dates: First submitted 2011-01-21; First posted 2011-01-24 (Estimated); Last update posted 2019-07-01 (Actual); Status verified 2013-07

CONDITIONS: Postmenopausal Symptoms; Hot Flashes
Keywords: Randomized Controlled Trial; Clinical Tria; Postmenopause; Hot-flashes; Quality of life; Physical Fitness
MeSH Terms: conditions — Hot Flashes | interventions — Physical Fitness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Increased Physical Activity (Experimental): Individually tailored training one hour, 2-3 sessions per week.
  Interventions: Behavioral: Physical activity intervention program
- Activity as usual ("Buisness as usual") (No Intervention)

INTERVENTIONS:
Behavioral: Physical activity intervention program — Individually tailored exercise programme (combination of pilates and aerobe training) with one hour activity sessions two-three times per week in 16 weeks.
  Other Names: Postmenoapsual symptoms; VO2-max; Physical fitness
  Arms: Increased Physical Activity

SUMMARY:
More than 60 % of women experience hot-flashes during postmenopausal and 20 % have serious symptoms. Use of combined estrogen/progesterone therapy reduces hot-flashes effectively. In 2001, results from the randomized controlled WHI-study (Womens Health Initiative) showed increased risk for breast cancer and hearth-disease among users of combined estrogen/progesterone therapy. This reduced the use of combined estrogen/progesterone therapy. Many women seek alternative treatment for hot-flashes. They are often told that physical activity can reduce intensity and frequency of hot-flashes. The evidence for this advice is sparse.

The primary hypothesis tested in the WHAT-study will be: Increased physical activity reduce frequency and intensity of hot-flushes among sedentary postmenopausal women with bothersome hot-flushes.

The WHAT-study is designed as a pragmatic randomized controlled clinical trial. To answer the primary hypothesis we will need approximately 500 participants. The logistic in a pragmatic trial of a complex intervention are complicated and we decided to first run a pilot study with 50 participants as a feasibility study. The pilot gives us opportunity to gain experience with possible problems like withdrawals and injuries.

DETAILED DESCRIPTION:
The WHAT study is a pragmatic randomized controlled trial with two parallel arms. The intervention is a 16 weeks individually tailored training programme with one hour physical activity 2-3 times per week. Women randomized to the control group are asked to keep physical activity at the same level as before the study.

Healthy postmenopausal women from Tromso will be recruited to the study by newspaper advertisements and media coverage. Interested women are asked to make a call. A staff member will ask about menopausal status, level of physical activity and diseases. Potential participants will receive a diary by mail and will be asked to record frequency and severity of hot-flashes, and duration of sleep at night for a period of 14 days. Women who return this diary will be asked to sign the informed consent and complete a questionnaire, before the fitness test. Baseline fitness is an important measure in this study. We will measure VO2-max (maximal oxygen consumption) as a proxy for fitness. Whether you are randomized to intervention or control group can influence the fitness test. The participants will therefore be randomized after the fitness test.

Randomization: Unit of Applied Clinical Research, Institute of Cancer Research and Molecular Medicine, Norwegian University of Science and Technology, Trondheim, Norway, will develop and administrate a web-based randomization system for the WHAT pilot study. The data base will be located at a server at the Medical Faculty at Norwegian University of Science and Technology in Trondheim. The following staff are authorized to randomize people in WHAT pilot study: Sameline Grimsgaard, Merethe Kumle, Sissel Andersen , Jorid Degerstrøm, Svein Arne Pettersen

In this pilot 50 women will be randomized either to intervention group (25 women) or control group (25 women).

Elements in the intervention: A physiotherapist will based on interview and physical examination make a plan for the 16 weeks physical activity programme for each participant. The program will start with Pilates classes and low intensity aerobic training (2-4 weeks). After this period, classes with moderate to high intensity aerobic training will be introduced. The aim of the intervention is to increase aerobic capacity with 10 % from baseline.

Both the intervention group and the control group will receive questionnaires at baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 6 months and 1 year after inclusion. We will run the test for physical fitness at baseline and 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal
* Natural or induced menopause
* > 12 months since last menstruation
* Severe hot flushes (frequency and intensity)
* Sedentary life style
* Motivated to increase level of physical activity

Exclusion Criteria:

* Current use of estrogen/progesterone treatment.
* Physical active (mean activity last six months
* More than 30 min per regularly exercise sessions at least once a week.
* Regular exercise sessions are defined as any planned physical activity (e.g., brisk walking, aerobics, jogging, bicycling, swimming, rowing, etc.) performed to increase physical fitness. BMI > 35 kg/m2, disease of illness that can hamper regular training.
* Current use of HT (systemic or plaster) during last 8 weeks

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in mean hot-flashes frequency and intensity (per 24/hours). | Baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks , 6 months and 1 year
  Potential participants receive a diary by mail and are asked to record frequency and severity of hot flashes and duration of sleep at night for a period of 14 subsequent days. During the study period the participants record frequency and intensity of hot flashes and duration of sleep at night for a period of 7 subsequent days at 4, 8, 12, 16 weeks and 6 months and one year.

SECONDARY OUTCOMES:
Quality of life measured with Women's Health Questionnaire (WHQ) 23 items. | Baseline, 16 weeks, 6 months, one year.
  We will measure quality of life with Women's Health Questionnaire. This is a self-administered questionnarie. A Norwegian version has been validated psychometric and linguistically.
Depressive symptoms are measured with Beck Depression Inventory -II (BDI-II) | Baseline, 16 weeks, 6 months
  The Beck Depression Inventory - Second Edition (BDI-II; Beck et al., 1996) is a 21-item self-report inventory designed to assess the presence and severity of depressive symptoms and is rated on a four-point Likert-type scale ranging from 0 to 3, reflecting the severity of each item. The BDI-II scores are classified as following: 0-13 minimal; 14-19 mild; 20-28 moderate; and 29-63 severe (Beck et al., 1996). A full description of the inventory including psychometric properties can be found in Steer, Ball, Ranieri, and Beck (1999).
Dysfunctional attitudes related to cognitive vulnerability to depression. | Baseline, 16 weeks, 6 months
  The Dysfunctional Attitude Scale (DAS)(Form A) (DAS; Weisman & Beck, 1978) is a 40-item self-report inventory to be rated along a seven-point Likert scale ranging from "totally agree" to "totally disagree", designed to assess the presence of dysfunctional attitudes that may relate to cognitive vulnerability to depression (Oliver & Baumgart, 1985). A full description including psychometric properties is provided by Chioqueta and Stiles (2004), Dobson and Breiter (1983) and Oliver and Baumgart (1985).
Increased physical fitness, measured as 10 % increase in VO2-max | Baseline, 16 weeks
  Physical fitness will be tested at the Regional Centre for Sport and Health, University of Tromsø, at baseline and after 16 weeks. VO2-max is used as a proxy for physical fitness.
Motivation for change in physical activity - Stages of Change | Baseline, 16 uker, 6 months and one year
  Permanent changes of behavior is difficult. We will use instruments from the Transtheoretical Model of Change, the Stages of Change short and long form to evaluate motivation for increased physical activity among the participants in the WHAT pilot study. The instrument might give valuable information about who a prone drop-out during study period.
Physical activity, motivation and experiences | Betwen 2nd and 16th week
  During the study period approximately 20 women (both from the intervention group and the control group) will be asked to participate i a qualitative study of physical activity, motivation and experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Sameline Grimsgaard, MD, PhD, Principal Investigator — University Hospital North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Troms, Norway